CLINICAL TRIAL: NCT06960070
Title: One-year Clinical Evaluation of Onlay Restorations Fabricated With Three Different Additive Manufacturing Resins in Endodontically Treated Teeth: A Prospective Study
Brief Title: Clinical Success of Onlays Fabricated With Different Types of Resin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Esra Cengiz Yanardag, Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025/364
Record Dates: First submitted 2025-04-18; First posted 2025-05-07 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Endodontically-Treated Teeth
Keywords: onlay; endodontically -reated teeth; indirect restoration; additively manufactured; hybrid resin
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Saremco print resin (Active Comparator)
  Interventions: Device: Saremco print resin
- Varseosmile Crownplus resin (Active Comparator)
  Interventions: Device: Varseosmile Crownplus resin
- Varseosmile TriniQ resin (Active Comparator)
  Interventions: Device: Varseosmile TriniQ resin

INTERVENTIONS:
Device: Saremco print resin — The teeth were restored with Saremco print resin via Asiga Max printer according to the manufacturer's instructions.
  Arms: Saremco print resin
Device: Varseosmile Crownplus resin — The teeth were restored with Varseosmile Crownplus resin via Asiga Max printer according to the manufacturer's instructions.
  Arms: Varseosmile Crownplus resin
Device: Varseosmile TriniQ resin — The teeth were restored with Varseosmile TriniQ resin via Asiga MAx printer according to the manufacturer' instructions
  Arms: Varseosmile TriniQ resin

SUMMARY:
Additive manufacturing, also referred to as "3D printing" or "rapid prototyping," is defined as the process of joining materials layer by layer to create an object based on 3D model data. In this method, a digital data set is first created on a computer (computer-aided design, CAD) and then transferred to a 3D printer. The designed object is produced by printing it in successive layers.

In contrast, in subtractive manufacturing, restorations are produced by milling homogeneous blocks based on computer-designed models. Compared to subtractive manufacturing technology, additive manufacturing allows for the production of more complex, detailed, and larger structures with much less material waste and without excessive use of force.

It is thought that additive manufacturing has the potential to overcome the disadvantages of subtractive manufacturing. Over the past decade, global sales of industrial and personal 3D printers, materials, and services have increased by more than 33% annually.

Due to its success in the production of surgical guides, temporary and permanent restorations, crowns and bridges, occlusal splints, frameworks, and orthodontic appliances, this technology has attracted significant interest in the field of dentistry.

Although additive manufacturing has started to be used as an alternative to subtractive manufacturing in many applications, there is still a lack of information regarding the chemical composition, mechanical, and physical properties of printable resins. Moreover, clinical data on the use of these resins in permanent restorations are quite limited.

Therefore, the aim of this study is to clinically evaluate and monitor for one year the performance of onlay restorations fabricated with three different resins of varying compositions in endodontically treated teeth.

ELIGIBILITY:
Inclusion Criteria:

* Molar teeth that have undergone root canal treatment
* Teeth with proximal defects located above the gingival margin
* Defects limited to the occlusal surface and a single adjacent surface
* Presence of an occlusal defect extending over one-third of the distance between the fissure and the cusp tip and involving one or more cusps
* Presence of an opposing tooth or a fixed prosthetic restoration against the tooth to be restored
* Presence of adjacent teeth next to the tooth to be restored

Exclusion Criteria:

* Fractured or cracked teeth
* Patients with temporomandibular joint disorders
* Patients with bruxism (teeth grinding)
* Molar teeth without an opposing tooth or fixed prosthetic restoration
* Molar teeth without adjacent teeth
* Vital teeth
* Patients with a history of allergy to the components of the resins

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2027-06-18 (Estimated)

PRIMARY OUTCOMES:
Clinical performance | Baseline- 6 months-12 months
  The clinical evaluation of restorations bonded to teeth will be performed at baseline, at 6 months, and at 12 months using the World Dental Federation (FDI) criteria which are divided into 3 main categories as functional, biological and esthetic properties. Each property is typically scored on a 1 to 5 scale:
  1. - Clinically excellent
  2. - Clinically good
  3. - Clinically sufficient
  4. - Clinically insufficient
  5. - Clinically poor

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Mersin University Faculty of Dentistry, Mersin, Mersin
  - Mersin University, Mersin, Mersin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code